CLINICAL TRIAL: NCT01215097
Title: A Randomized, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Study of BI 1356 Over 24 Weeks in T2D Patients With Insufficient Glycaemic Control Despite Metformin Therapy
Brief Title: Efficacy and Safety Study of Linagliptin (5 mg Administered Orally Once Daily) Over 24 Weeks in Type 2 Diabetic Patients With Insufficient Glycaemic Control Despite Metformin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.65
Record Dates: First submitted 2010-09-28; First posted 2010-10-06 (Estimated); Results first posted 2013-06-03 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin (Experimental): once a day
  Interventions: Drug: Linagliptin
- placebo (Placebo Comparator): once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Linagliptin — once a day
  Arms: Linagliptin
Drug: placebo — once a day
  Arms: placebo

SUMMARY:
In this randomised, double-blind, parallel group trial, the safety and efficacy of 5 mg of Linagliptin administered orally once daily will be compared with a placebo after 24 weeks of treatment as add-on therapy to metformin in patients with type 2 diabetes and insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Male and female patients with a diagnosis of type 2 diabetes mellitus and previously treated with metformin alone, or with metformin and not more than one other oral antidiabetic drug (antidiabetic therapy has to be unchanged for 6 weeks prior to informed consent and patients should receive standard diet and exercise counseling) A dose of >/=1500 mg/day metformin is required for inclusion into the trial. The dosage needs to be stable for at least 8 weeks before randomisation. Patients with a total daily dose of less than 1500 mg metformin will only be included; if the investigator has documented them to be on their maximum tolerated dose (also in this case the 8 week time interval will apply for a stable dose).
2. Diagnosis of type 2 diabetes prior to informed consent
3. Glycosylated haemoglobin A1 (HbA1c) at Visit 1a (Screening):

   For patients undergoing wash out of previous medication: HbA1c =7.0 to =9.5% For patients not undergoing wash-out of previous medication: HbA1c =7.0 to =10.0%
4. Glycosylated haemoglobin A1 (HbA1c) =7.0 to =10.0% at Visit 2 (Start of Run-in)
5. Age = 18 and < 80 years at Visit 1a (Screening)
6. BMI (Body Mass Index) = 45 kg/m2 at Visit 1a (Screening)
7. Signed and dated written informed consent by date of Visit 1a in accordance with GCP and local legislation

Exclusion criteria:

1. Myocardial infarction, stroke or TIA within 6 months prior to informed consent
2. Impaired hepatic function, defined by serum levels of either Alanine transaminase,Aspartate transaminase, or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at Visit 1a
3. Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during wash-out / placebo run-in and confirmed by a second measurement (not on the same day).
4. Known hypersensitivity or allergy to the investigational product or its excipients or metformin or placebo
5. Treatment with rosiglitazone or pioglitazone within 3 months prior to informed consent
6. Treatment with an injectable Glucagon-like peptide- 1 (GLP-1) analogue (e.g. exenatide) , Dipeptidyl-Peptidase 4 (DPP-IV) inhibitor within 3 months prior to informed consent
7. Treatment with insulin within 3 months prior to informed consent
8. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat, rimonabant) within 3 months prior to informed consent.
9. Alcohol abuse within the 3 months prior to informed consent that would interfere with trial participation or drug abuse
10. Participation in another trial with an investigational drug within 2 months prior to informed consent
11. Pre-menopausal women (last menstruation =1 year prior to informed consent) who:

    * are nursing or pregnant,
    * or are of child-bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include transdermal patch, intra-uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner. No exception will be made.
12. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent.
13. Renal failure or renal impairment (serum creatinine =1.5 mg/dl as determined at Visit 1a)
14. Dehydration by clinical judgement of the investigator
15. Unstable or acute congestive heart failure
16. Acute or chronic metabolic acidosis (present in patient history)
17. Hereditary galactose intolerance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (19):
- China (15):
  - 1218.65.86007 Boehringer Ingelheim Investigational Site, Beijing
  - 1218.65.86011 Boehringer Ingelheim Investigational Site, Chongqing
  - 1218.65.86008 Boehringer Ingelheim Investigational Site, Dalian
  - 1218.65.86010 Boehringer Ingelheim Investigational Site, Fuzhou
  - 1218.65.86014 Boehringer Ingelheim Investigational Site, Hangzhou
  - 1218.65.86005 Boehringer Ingelheim Investigational Site, Hefei
  - 1218.65.86006 Boehringer Ingelheim Investigational Site, Hefei
  - 1218.65.86012 Boehringer Ingelheim Investigational Site, Nanjing
  - 1218.65.86001 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.65.86002 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.65.86003 Boehringer Ingelheim Investigational Site, Shanghai
  - 1218.65.86004 Boehringer Ingelheim Investigational Site, Suzhou
  - 1218.65.86015 Boehringer Ingelheim Investigational Site, Wenzhou
  - 1218.65.86009 Boehringer Ingelheim Investigational Site, Wuhan
  - 1218.65.86013 Boehringer Ingelheim Investigational Site, Yangzhou
- Malaysia (2):
  - 1218.65.60002 Boehringer Ingelheim Investigational Site, Johor Bahru
  - 1218.65.60001 Boehringer Ingelheim Investigational Site, Kelantan
- Philippines (2):
  - 1218.65.63001 Boehringer Ingelheim Investigational Site, Marikina City
  - 1218.65.63002 Boehringer Ingelheim Investigational Site, San Juan City

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 614 patients were screened in 19 centres in China, Malaysia,and Philippines.A total of 306 patients were randomised in a 1:2 ratio to receive either placebo (101 patients) or linagliptin 5 mg (205 patients) in addition to metformin.
Groups:
- Placebo: Placebo
- Linagliptin 5mg: Linagliptin 5mg, once daily tablets, oral
Period: Overall Study
Arm/Group | Placebo | Linagliptin 5mg
Started | 100 (Patients who are randomised and treated with placebo. 1 patient was not treated then not included.) | 205 (Patients who are randomised and treated with linagliptin.)
Completed | 88 | 191
Not Completed | 12 | 14
Not completed — Adverse Event | 1 | 3
Not completed — Protocol Violation | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 6 | 3
Not completed — Lack of Efficacy | 0 | 3
Not completed — patient's refusal to come | 2 | 2
Not completed — patient's private reason | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Linagliptin 5mg | Total
Number analyzed (Participants) | 100 | 205 | 305
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (8.7) | 55.1 (10.7) | 55.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 103 | 153
  Male | 50 | 102 | 152
BMI [Mean (Standard Deviation); unit: kg/m^2] — Baseline body mass index (BMI)
  kg/m^2 | 25.8 (4.0) | 25.5 (3.9) | 25.6 (4.0)
Baseline HbA1c [Mean (Standard Deviation); unit: %] — Baseline HbA1c
  % | 8.00 (0.80) | 7.99 (0.83) | 7.99 (0.82)
Baseline fasting plasma glucose [Mean (Standard Deviation); unit: mg/dL] — Baseline fasting plasma glucose
  mg/dL | 157.7 (36.8) | 160.5 (40.1) | 159.6 (39.0)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline at Week 24
Description: Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and at week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Percent | -0.14 (0.07) | -0.66 (0.05)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.52, 95% CI [-0.70 to -0.34], Standard Error of Mean 0.09

2. Secondary Outcome: HbA1c Change From Baseline at Week 6
Description: Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and at week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Percent | -0.02 (0.052) | -0.455 (0.037)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.433, 95% CI 2-sided [-0.555 to -0.311], Standard Error of Mean 0.062

3. Secondary Outcome: HbA1c Change From Baseline at Week 12
Description: Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Percent | -0.062 (0.068) | -0.653 (0.048)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.591, 95% CI [-0.752 to -0.43], Standard Error of Mean 0.082

4. Secondary Outcome: HbA1c Change From Baseline at Week 18
Description: Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and at week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Percent | -0.119 (0.073) | -0.645 (0.052)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.53, 95% CI [-0.70 to -0.35], Standard Error of Mean 0.09

5. Secondary Outcome: HbA1c Change From Baseline at Week 24(Chinese Only)
Description: Means are treatment adjusted for baseline HbA1c and previous anti-diabetic medication.
Time Frame: Baseline and at 24 weeks
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available (Chinese only). Last observation carried forward (LOCF) was used as the imputation rule.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 77 | 182
Percent | -0.16 (0.08) | -0.68 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -0.52, 95% CI [-0.71 to -0.32], Standard Error of Mean 0.1

6. Secondary Outcome: FPG Change From Baseline at Week 24
Description: Means are treatment adjusted for baseline fasting plasma glucose (FPG) and previous anti-diabetic medication.
Time Frame: Baseline and at week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
mg/dL | -1.1 (3.5) | -10.7 (2.5)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0233, ANCOVA; Adjusted mean difference = -9.6, 95% CI [-17.8 to -1.3], Standard Error of Mean 4.2

7. Secondary Outcome: FPG Change From Baseline at Week 6
Description: Means are treatment adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and at week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
mg/dL | 5.3 (2.8) | -16.8 (2.0)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Adjusted mean difference = -22.1, 95% CI [-28.7 to -15.6], Standard Error of Mean 3.3

8. Secondary Outcome: FPG Change From Baseline at Week 12
Description: Means are treatment adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and at week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
mg/dL | -4.5 (3.0) | -14.7 (2.1)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0050, ANCOVA; Adjusted mean difference = -10.2, 95% CI [-17.3 to -3.1], Standard Error of Mean 3.6

9. Secondary Outcome: FPG Change From Baseline at Week 18
Description: Means are treatment adjusted for baseline FPG and previous anti-diabetic medication.
Time Frame: Baseline and at week 18
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
mg/dL | -1.9 (3.4) | -13.4 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Test type: Superiority or Other; p = 0.0044, ANCOVA; Adjusted mean difference = -11.5, 95% CI [-19.5 to -3.6], Standard Error of Mean 4.0

10. Secondary Outcome: Number of Patients With HbA1c < 7.0%
Description: Number of patients with HbA1c < 7.0% at week 24
Time Frame: baseline and at week 24
Population: The Full Analysis Set (FAS) included all treated and randomised patients with a baseline and at least one on-treatment HbA1c measurement available. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Participants | 14 | 82

11. Secondary Outcome: Number of Patients With HbA1c < 7.0% at Week 24 With Baseline HbA1c >= 7.0%.
Description: Number of patients with HbA1c < 7.0% at week 24 with baseline HbA1c >= 7.0%.
Time Frame: baseline and at week 24
Population: This population includes the FAS with baseline HbA1c >= 7.0%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 89 | 185
Participants | 9 | 69
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Comparison by odds ratio for the patients with a baseline HbA1c >=7.0%; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 6.243, 95% CI [2.831 to 13.769]

12. Secondary Outcome: Number of Patients With HbA1c < 6.5%
Description: Number of patients with HbA1c < 6.5% at week 24
Time Frame: baseline and at week 24
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Participants | 4 | 26

13. Secondary Outcome: Number of Patients With HbA1c < 6.5% at Week 24 With Baseline HbA1c >= 6.5%.
Description: Number of patients with HbA1c < 6.5% at week 24 with baseline HbA1c >= 6.5%.
Time Frame: baseline and at week 24
Population: This population includes the FAS with baseline HbA1c >= 6.5%. Non-completers were considered as failure imputation (NCF).
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 96 | 202
Participants | 3 | 26
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Comparison by odds ratio for the patients with a baseline HbA1c >= 6.5%; Test type: Superiority or Other; p = 0.0129, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 4.97, 95% CI [1.404 to 17.592]

14. Secondary Outcome: Number With HbA1c at Least Lowering 0.5%
Description: Number with HbA1c at least 0.5% lowering from baseline at week 24
Time Frame: baseline and at week 24
Population: as for outcome 10
Measure: Number; unit: Participants
Arm/Group | Placebo | Linagliptin 5mg
Number analyzed (Participants) | 97 | 203
Participants | 33 | 120
Statistical Analysis 1: Comparison: Placebo vs Linagliptin 5mg; Comparison by odds ratio for the patients with HbA1c at least lowering 0.5% from baseline; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The odds-ratio is based on a logistic regression model including baseline HbA1c and previous antidiabetic medication; Odds Ratio (OR) = 3.054, 95% CI [1.799 to 5.185]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Placebo | Linagliptin 5mg
Serious Adverse Events (participants affected / at risk) | 2/100 | 4/205
Other Adverse Events (participants affected / at risk) | 13/100 | 29/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Linagliptin 5mg (N=205)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Linagliptin 5mg (N=205)
Upper respiratory tract infection (Infections and infestations) | 3 | 3
Nasopharyngitis (Infections and infestations) | 1 | 5
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 10
Diarrhoea (Gastrointestinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes